CLINICAL TRIAL: NCT05640648
Title: Human-centered Design and Communities of Practice to Improve Delivery of Home-based Tuberculosis Contact Investigation in Uganda
Brief Title: Human-centered Design and Communities of Practice to Improve Home-based Tuberculosis Contact Investigation in Uganda
Acronym: HCD-CoP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Screening
Other Study IDs: R01AI104824 (NIH); 5R01AI104824 (NIH); R01AI104824 (NIH); 2000023199 (Other: Yale IRB)
Record Dates: First submitted 2022-11-16; First posted 2022-12-07 (Actual); Results first posted 2025-03-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Tuberculosis; Tuberculosis, Pulmonary
MeSH Terms: conditions — Tuberculosis; Tuberculosis, Pulmonary

STUDY DESIGN:
Intervention Model Description: The investigators will conduct a stepped-wedge, cluster-randomized implementation trial with nested mixed-methods evaluations of fidelity and context and health economic analyses. The stepped-wedge trial will include six transition steps in a complete (also known as closed) design, providing a 1:1 ratio of time periods allocated to the pre-implementation standard strategy and the post-implementation user-centered strategy.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Blinding of the assigned intervention is not feasible with the stepped-wedge cluster randomized implementation trial design, because interventions are implemented at the health-facility level and all health facilities receive the standard strategy followed by the enhanced, user-centered strategy. Community Health Workers will collect all data, and adjudicate all outcomes, except TB diagnoses and treatments initiated which will be collected from on-site National TB and Leprosy Programme registers. Where possible, the investigators and study staff, except for the statistician and data manager, will be blinded to any aggregated analyses of TB outcomes by study period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Implementation Strategy Period (Active Comparator): During the standard implementation strategy period, CHWs at all sites will receive the standard TB program training on TB contact investigation and supportive supervision from the on-site National TB Program focal person.
  Interventions: Behavioral: Standard Implementation Strategy
- Enhanced Contact Investigation Intervention Period (Experimental): The enhanced contact investigation strategy includes 4 implementation facilitation tools and 3 continuous quality improvement techniques and will be delivered as a branded package named for an inspirational Luganda phrase that is translated as "We are together with you." Implementation facilitation tools include 1) a TB education pamphlet, 2) a contact identification algorithm, 3) an instructional video on sputum collection, and 4) community health riders who transport clients, community health workers, and sputum samples by motorcycle. The continuous quality improvement techniques delivered as the community of practice package include 1) community of practice meetings, 2) audit and feedback reports and 3) a group chat application.
  Interventions: Behavioral: User-Centered Implementation Strategy

INTERVENTIONS:
Behavioral: User-Centered Implementation Strategy — 1. 4 participant-facing components: 1a) TB education pamphlet helps index TB persons disclose the need for household screening to contacts. 1b) Contact identification algorithm helps CHWs and index TB persons accurately enumerate contacts. 1c) Sputum collection video instructs contacts to expectorate good-quality sputum. 1d) Community Health Riders transport CHWs, index persons with TB, and contacts by motorcycle taxi, and collect and transport sputum.
  2. 3 community health-worker-facing components: a) Weekly CHW meetings create communities of practice (CoP), professionals organized for peer support and systematic learning. Meetings involve problem solving, review of audit and feedback reports, and didactics on TB care, among other activities. 2b) Audit and feedback reports on contact investigation performance indicators weekly (individual CHW) and monthly (health facility). 2c) A group-chat application facilitates peer support among CHWs.
  Other Names: Enhanced Contact Investigation Implementation Strategy
  Arms: Enhanced Contact Investigation Intervention Period
Behavioral: Standard Implementation Strategy — Once an eligible TB patient agrees to participate, CHWs will visit the patient to assess the eligibility of close contacts to participate. For eligible contacts who agree to participate, the CHW will perform TB symptom screening and arrange subsequent microbiologic, clinical, and/or radiographic evaluation. Those screening TB symptom-positive will be asked to expectorate a sputum sample, unless under age 5. If under age 5 or unable to produce sputum, contacts will be referred to the health centre for evaluation. A CHW will transport sputum samples to the health-centre laboratory for microbiologic evaluation and later report the test results back to the contact. During the standard implementation strategy period, CHWs at all sites will receive the standard TB program training on TB contact investigation and supportive supervision from the on-site National TB Program focal person.
  Other Names: Usual Implementation Strategy
  Arms: Standard Implementation Strategy Period

SUMMARY:
In a previous randomized control trial, the investigators identified gaps in the implementation of tuberculosis (TB) contact investigation at multiple levels of the service delivery cascade. Drawing on prior experiences, the investigators have recently developed a novel strategy to enhance the implementation of routine contact investigation procedures. This user-centered implementation strategy was created through serial prototyping guided by human-centered design (HCD) and employs communities of practice (CoP) as an adjunctive adaptation and sustainment strategy. The investigators are now conducting a stepped-wedge, cluster-randomized implementation trial in 12 study sites in Uganda to determine if the resulting user-centered implementation strategy enhances the delivery of TB contact investigation and other implementation outcomes, and also improves health outcomes.

DETAILED DESCRIPTION:
The trial has 3 major aims: (1) to compare the implementation, effectiveness, and public health impact of TB contact investigation delivered via an enhanced, "user-centered" implementation strategy versus a standard implementation strategy in a stepped-wedge, cluster-randomized implementation trial; (2) to identify processes and contextual factors that influence the implementation, effectiveness, and public health impact of the enhanced delivery strategy for TB contact investigation; and (3) to compare the costs and epidemiological impact of the enhanced and standard implementation strategies for TB contact investigation. The enhanced, user-centered strategy will employ two major components: a) a branded, participant-centered strategy consisting of implementation facilitation tools previously developed using human-centered design; and b) Communities of Practice, a community-health worker-centered, continuous quality improvement strategy. The goal is to improve the delivery of standard TB contact investigation following Uganda National TB & Leprosy Programme guidelines. The investigators hypothesize that the enhanced, user-centered strategy will result in a greater proportion of close contacts completing TB evaluation than the standard strategy. They further hypothesize that successful implementation will be deemed feasible, acceptable, and appropriate by patients and CHWs and that it will increase self-efficacy and perceived social support among CHWs. Finally, the investigators hypothesize that models evaluating the impact of the user-centered strategy when delivered nationwide will find it cost-effective and able to reduce national TB incidence over a 10-year horizon.

ELIGIBILITY:
Health centre inclusion criteria:

1. Reporting ≥12 index TB cases per month to the national TB program,
2. Located outside the borders of but ≤180 km from Kampala District

Health centre exclusion criteria:

1) Administrators of the health centre do not agree to participate in the study

Individual inclusion criteria for index persons with TB (also known as index TB patients or TB cases):

1. Being an adult or child recorded as a new TB case in the on-site National TB and Leprosy Programme TB treatment register, and
2. Residing ≤40 km from the enrolling health centre,

Individual exclusion criteria for index persons with TB :

1. Lacking the capacity to consent to contact investigation,
2. Lacking close contacts,
3. Having possible or confirmed drug-resistant TB,
4. Previously received TB contact investigation within the last 2 months, and
5. Not agreeing to refer close contacts for contact investigation.

Inclusion criteria for close contacts:

1) Being an adult or child reporting ≥12 cumulative hours with the TB patient inside an enclosed space within the previous 3 months,

Exclusion criteria for close contacts:

1. Lacking the capacity to consent to contact investigation,
2. Currently taking treatment for active TB, and
3. Not agreeing to participate in contact investigation.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10477 (Actual)
Dates: Start 2022-03-07 (Actual); Primary Completion 2023-10-26 (Actual); Study Completion 2023-10-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J. Lucian Davis, MD, Principal Investigator — Yale School of Public Health
Locations (1):
- Uganda Tuberculosis Implementation Research Consortium, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication upon request
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: After primary trial results are published
Access Criteria: Upon request to the PI

REFERENCES:
- [Derived] Katamba A, Gupta AJ, Turimumahoro P, Ochom E, Ggita JM, Nakasendwa S, Nanziri L, Musinguzi J, Hennein R, Sekadde M, Hanrahan C, Byaruhanga R, Yoeli E, Turyahabwe S, Cattamanchi A, Dowdy DW, Haberer JE, Armstrong-Hough M, Kiwanuka N, Davis JL. A user-centred implementation strategy for tuberculosis contact investigation in Uganda: protocol for a stepped-wedge, cluster-randomised trial. BMC Public Health. 2023 Aug 17;23(1):1568. doi: 10.1186/s12889-023-16510-0. PMID 37592314
- [Derived] Katamba A, Gupta AJ, Turimumahoro P, Ochom E, Ggita JM, Nakasendwa S, Nanziri L, Musinguzi J, Hennein R, Sekadde M, Hanrahan C, Byaruhanga R, Yoeli E, Turyahabwe S, Cattamanchi A, Dowdy DW, Haberer JE, Armstrong-Hough M, Kiwanuka N, Davis JL. A user-centred implementation strategy for tuberculosis contact investigation in Uganda: Protocol for a stepped-wedge, cluster-randomised trial. Res Sq [Preprint]. 2023 Jul 6:rs.3.rs-3121275. doi: 10.21203/rs.3.rs-3121275/v1. PMID 37461631

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In this stepped-wedge, cluster-randomized trial, 12 health facilities progress from Standard Contact Investigation [Control] to User-centered Contact Investigation [Intervention] in 6 clusters of randomly assigned pairs that cross over one cluster at a time [Sequences] at randomly assigned 8-week intervals [Periods]. All clusters start in Standard for 8 weeks, then 1 cluster crosses over to User-centered every 8 weeks for 48 weeks, and finally all clusters are in User-centered for 8 weeks.
Units Other Than Participants: Pairs of Health Facilities
Groups:
- Standard Contact Investigation [Control]: Sequence 1 [2 Health Facilities]: Cluster 1: 8 weeks of standard, then 8 weeks of transition, then 48 weeks of user-centered
  ----------------- Standard contact investigation consists of 1) evidence-based procedures for TB contact investigation, introduced with 2) a standard implementation strategy.
  1. Standard contact investigation:
     1. Once an eligible TB patient agrees to participate, CHWs will visit the patient to assess the eligibility of close contacts to participate.
     2. For eligible contacts who agree to participate, the CHW will perform TB symptom screening and arrange subsequent microbiologic, clinical, and/or radiographic evaluation. c) Those screening TB symptom-positive will be asked to expectorate a sputum sample, unless under age 5. If under age 5 or unable to produce sputum, contacts will be referred to the health centre for evaluation. A CHW will transport sputum samples to the health-centre laboratory for microbiologic evaluation and later report the test results back to the contact.
  2. Standard Implementation Strategy:
  CHWs at all sites will receive the standard TB program training on TB contact investigation and supportive supervision from the on-site National TB Program focal person.
- User-centered Contact Investigation [Intervention]: Sequence 1 [2 Health Facilities]: Cluster 1: 8 weeks of standard, then 8 weeks of transition, then 48 weeks of user-centered
  ----------------- User-centered Contact Investigation includes 4 client-facing adaptations of standard contact investigation and 3 CHW-facing implementation strategies
  1. Client-centered adaptations of contact investigation delivered as a branded package called Tuli Wamu Nawe: Four novel tools
     1. TB education pamphlet to help index TB persons disclose the need for TB screening to close contacts.
     2. Contact identification algorithm to help CHWs and index TB persons accurately enumerate contacts.
     3. Sputum collection video to instruct contacts to expectorate good-quality sputum.
     4. Community Health Riders to transport CHWs, index persons with TB, and contacts by motorcycle taxi, and collect and transport sputum.
  2. CHW-centered Implementation Strategy: Three components
     1. Weekly CHW meetings to create communities of practice (CoP), which consist of professionals organized for peer support and systematic learning.
     2. Audit and feedback reports on contact investigation performance indicators delivered weekly (individual CHW) and monthly (health facility).
     3. A group-chat application to facilitate peer support among CHWs.
- Standard Contact Investigation [Control]: Sequence 2 [2 Health Facilities]: Cluster 2: 16 weeks of standard, then 8 weeks of transition, then 40 weeks of user-centered
  ----------------- Standard contact investigation consists of 1) evidence-based procedures for TB contact investigation, introduced with 2) a standard implementation strategy.
  1. Standard contact investigation:
     1. Once an eligible TB patient agrees to participate, CHWs will visit the patient to assess the eligibility of close contacts to participate.
     2. For eligible contacts who agree to participate, the CHW will perform TB symptom screening and arrange subsequent microbiologic, clinical, and/or radiographic evaluation. c) Those screening TB symptom-positive will be asked to expectorate a sputum sample, unless under age 5. If under age 5 or unable to produce sputum, contacts will be referred to the health centre for evaluation. A CHW will transport sputum samples to the health-centre laboratory for microbiologic evaluation and later report the test results back to the contact.
  2. Standard Implementation Strategy:
  CHWs at all sites will receive the standard TB program training on TB contact investigation and supportive supervision from the on-site National TB Program focal person.
- User-centered Contact Investigation [Intervention]: Sequence 2 [2 Health Facilities]: Cluster 2: 16 weeks of standard, then 8 weeks of transition, then 40 weeks of user-centered
  ----------------- User-centered Contact Investigation includes 4 client-facing adaptations of standard contact investigation and 3 CHW-facing implementation strategies
  1. Client-centered adaptations of contact investigation delivered as a branded package called Tuli Wamu Nawe: Four novel tools
     1. TB education pamphlet to help index TB persons disclose the need for TB screening to close contacts.
     2. Contact identification algorithm to help CHWs and index TB persons accurately enumerate contacts.
     3. Sputum collection video to instruct contacts to expectorate good-quality sputum.
     4. Community Health Riders to transport CHWs, index persons with TB, and contacts by motorcycle taxi, and collect and transport sputum.
  2. CHW-centered Implementation Strategy: Three components
     1. Weekly CHW meetings to create communities of practice (CoP), which consist of professionals organized for peer support and systematic learning.
     2. Audit and feedback reports on contact investigation performance indicators delivered weekly (individual CHW) and monthly (health facility).
     3. A group-chat application to facilitate peer support among CHWs.
- Standard Contact Investigation [Control]: Sequence 3 [2 Health Facilities]: Cluster 3: 24 weeks of standard, then 8 weeks of transition, then 32 weeks of user-centered
  ----------------- Standard contact investigation consists of 1) evidence-based procedures for TB contact investigation, introduced with 2) a standard implementation strategy.
  1. Standard contact investigation:
     1. Once an eligible TB patient agrees to participate, CHWs will visit the patient to assess the eligibility of close contacts to participate.
     2. For eligible contacts who agree to participate, the CHW will perform TB symptom screening and arrange subsequent microbiologic, clinical, and/or radiographic evaluation. c) Those screening TB symptom-positive will be asked to expectorate a sputum sample, unless under age 5. If under age 5 or unable to produce sputum, contacts will be referred to the health centre for evaluation. A CHW will transport sputum samples to the health-centre laboratory for microbiologic evaluation and later report the test results back to the contact.
  2. Standard Implementation Strategy:
  CHWs at all sites will receive the standard TB program training on TB contact investigation and supportive supervision from the on-site National TB Program focal person.
- User-centered Contact Investigation [Intervention]: Sequence 3 [2 Health Facilities]: Cluster 3: 24 weeks of standard, then 8 weeks of transition, then 36 weeks of user-centered
  ----------------- User-centered Contact Investigation includes 4 client-facing adaptations of standard contact investigation and 3 CHW-facing implementation strategies
  1. Client-centered adaptations of contact investigation delivered as a branded package called Tuli Wamu Nawe: Four novel tools
     1. TB education pamphlet to help index TB persons disclose the need for TB screening to close contacts.
     2. Contact identification algorithm to help CHWs and index TB persons accurately enumerate contacts.
     3. Sputum collection video to instruct contacts to expectorate good-quality sputum.
     4. Community Health Riders to transport CHWs, index persons with TB, and contacts by motorcycle taxi, and collect and transport sputum.
  2. CHW-centered Implementation Strategy: Three components
     1. Weekly CHW meetings to create communities of practice (CoP), which consist of professionals organized for peer support and systematic learning.
     2. Audit and feedback reports on contact investigation performance indicators delivered weekly (individual CHW) and monthly (health facility).
     3. A group-chat application to facilitate peer support among CHWs.
- Standard Contact Investigation [Control]: Sequence 4 [2 Health Facilities]: Cluster 4: 32 weeks of standard, then 8 weeks of transition, then 24 weeks of user-centered
  ----------------- Standard contact investigation consists of 1) evidence-based procedures for TB contact investigation, introduced with 2) a standard implementation strategy.
  1. Standard contact investigation:
     1. Once an eligible TB patient agrees to participate, CHWs will visit the patient to assess the eligibility of close contacts to participate.
     2. For eligible contacts who agree to participate, the CHW will perform TB symptom screening and arrange subsequent microbiologic, clinical, and/or radiographic evaluation. c) Those screening TB symptom-positive will be asked to expectorate a sputum sample, unless under age 5. If under age 5 or unable to produce sputum, contacts will be referred to the health centre for evaluation. A CHW will transport sputum samples to the health-centre laboratory for microbiologic evaluation and later report the test results back to the contact.
  2. Standard Implementation Strategy:
  CHWs at all sites will receive the standard TB program training on TB contact investigation and supportive supervision from the on-site National TB Program focal person.
- User-centered Contact Investigation [Intervention]: Sequence 4 [2 Health Facilities]: Cluster 4: 32 weeks of standard, then 8 weeks of transition, then 24 weeks of user-centered
  ----------------- User-centered Contact Investigation includes 4 client-facing adaptations of standard contact investigation and 3 CHW-facing implementation strategies
  1. Client-centered adaptations of contact investigation delivered as a branded package called Tuli Wamu Nawe: Four novel tools
     1. TB education pamphlet to help index TB persons disclose the need for TB screening to close contacts.
     2. Contact identification algorithm to help CHWs and index TB persons accurately enumerate contacts.
     3. Sputum collection video to instruct contacts to expectorate good-quality sputum.
     4. Community Health Riders to transport CHWs, index persons with TB, and contacts by motorcycle taxi, and collect and transport sputum.
  2. CHW-centered Implementation Strategy: Three components
     1. Weekly CHW meetings to create communities of practice (CoP), which consist of professionals organized for peer support and systematic learning.
     2. Audit and feedback reports on contact investigation performance indicators delivered weekly (individual CHW) and monthly (health facility).
     3. A group-chat application to facilitate peer support among CHWs.
- Standard Contact Investigation [Control]: Sequence 5 [2 Health Facilities]: Cluster 5: 40 weeks of standard, then 8 weeks of transition, then 16 weeks of user-centered
  ----------------- Standard contact investigation consists of 1) evidence-based procedures for TB contact investigation, introduced with 2) a standard implementation strategy.
  1. Standard contact investigation:
     1. Once an eligible TB patient agrees to participate, CHWs will visit the patient to assess the eligibility of close contacts to participate.
     2. For eligible contacts who agree to participate, the CHW will perform TB symptom screening and arrange subsequent microbiologic, clinical, and/or radiographic evaluation. c) Those screening TB symptom-positive will be asked to expectorate a sputum sample, unless under age 5. If under age 5 or unable to produce sputum, contacts will be referred to the health centre for evaluation. A CHW will transport sputum samples to the health-centre laboratory for microbiologic evaluation and later report the test results back to the contact.
  2. Standard Implementation Strategy:
  CHWs at all sites will receive the standard TB program training on TB contact investigation and supportive supervision from the on-site National TB Program focal person.
- User-centered Contact Investigation [Intervention]: Sequence 5 [2 Health Facilities]: Cluster 5: 40 weeks of standard, then 8 weeks of transition, then 16 weeks of user-centered
  ----------------- User-centered Contact Investigation includes 4 client-facing adaptations of standard contact investigation and 3 CHW-facing implementation strategies
  1. Client-centered adaptations of contact investigation delivered as a branded package called Tuli Wamu Nawe: Four novel tools
     1. TB education pamphlet to help index TB persons disclose the need for TB screening to close contacts.
     2. Contact identification algorithm to help CHWs and index TB persons accurately enumerate contacts.
     3. Sputum collection video to instruct contacts to expectorate good-quality sputum.
     4. Community Health Riders to transport CHWs, index persons with TB, and contacts by motorcycle taxi, and collect and transport sputum.
  2. CHW-centered Implementation Strategy: Three components
     1. Weekly CHW meetings to create communities of practice (CoP), which consist of professionals organized for peer support and systematic learning.
     2. Audit and feedback reports on contact investigation performance indicators delivered weekly (individual CHW) and monthly (health facility).
     3. A group-chat application to facilitate peer support among CHWs.
- Standard Contact Investigation [Control]: Sequence 6 [2 Health Facilities]: Cluster 6: 48 weeks of standard, then 8 weeks of transition, then 8 weeks of user-centered
  ----------------- Standard contact investigation consists of 1) evidence-based procedures for TB contact investigation, introduced with 2) a standard implementation strategy.
  1. Standard contact investigation:
     1. Once an eligible TB patient agrees to participate, CHWs will visit the patient to assess the eligibility of close contacts to participate.
     2. For eligible contacts who agree to participate, the CHW will perform TB symptom screening and arrange subsequent microbiologic, clinical, and/or radiographic evaluation. c) Those screening TB symptom-positive will be asked to expectorate a sputum sample, unless under age 5. If under age 5 or unable to produce sputum, contacts will be referred to the health centre for evaluation. A CHW will transport sputum samples to the health-centre laboratory for microbiologic evaluation and later report the test results back to the contact.
  2. Standard Implementation Strategy:
  CHWs at all sites will receive the standard TB program training on TB contact investigation and supportive supervision from the on-site National TB Program focal person.
- User-centered Contact Investigation [Intervention]: Sequence 6 [2 Health Facilities]: Cluster 6: 48 weeks of standard, then 8 weeks of transition, then 8 weeks of user-centered
  ----------------- User-centered Contact Investigation includes 4 client-facing adaptations of standard contact investigation and 3 CHW-facing implementation strategies
  1. Client-centered adaptations of contact investigation delivered as a branded package called Tuli Wamu Nawe: Four novel tools
     1. TB education pamphlet to help index TB persons disclose the need for TB screening to close contacts.
     2. Contact identification algorithm to help CHWs and index TB persons accurately enumerate contacts.
     3. Sputum collection video to instruct contacts to expectorate good-quality sputum.
     4. Community Health Riders to transport CHWs, index persons with TB, and contacts by motorcycle taxi, and collect and transport sputum.
  2. CHW-centered Implementation Strategy: Three components
     1. Weekly CHW meetings to create communities of practice (CoP), which consist of professionals organized for peer support and systematic learning.
     2. Audit and feedback reports on contact investigation performance indicators delivered weekly (individual CHW) and monthly (health facility).
     3. A group-chat application to facilitate peer support among CHWs.
Period: Period 1 (Weeks 1-8)
Arm/Group | Standard Contact Investigation [Control]: Sequence 1 [2 Health Facilities] | User-centered Contact Investigation [Intervention]: Sequence 1 [2 Health Facilities] | Standard Contact Investigation [Control]: Sequence 2 [2 Health Facilities] | User-centered Contact Investigation [Intervention]: Sequence 2 [2 Health Facilities] | Standard Contact Investigation [Control]: Sequence 3 [2 Health Facilities] | User-centered Contact Investigation [Intervention]: Sequence 3 [2 Health Facilities] | Standard Contact Investigation [Control]: Sequence 4 [2 Health Facilities] | User-centered Contact Investigation [Intervention]: Sequence 4 [2 Health Facilities] | Standard Contact Investigation [Control]: Sequence 5 [2 Health Facilities] | User-centered Contact Investigation [Intervention]: Sequence 5 [2 Health Facilities] | Standard Contact Investigation [Control]: Sequence 6 [2 Health Facilities] | User-centered Contact Investigation [Intervention]: Sequence 6 [2 Health Facilities]
Started | 85; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities (In a stepped-wedge trial, enrollment is zero by design for certain sequences in certain periods.) | 297; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities (In a stepped-wedge trial, enrollment is zero by design for certain sequences in certain periods.) | 111; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities (In a stepped-wedge trial, enrollment is zero by design for certain sequences in certain periods.) | 134; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities (In a stepped-wedge trial, enrollment is zero by design for certain sequences in certain periods.) | 110; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities (In a stepped-wedge trial, enrollment is zero by design for certain sequences in certain periods.) | 176; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities (In a stepped-wedge trial, enrollment is zero by design for certain sequences in certain periods.)
Index Participants (Index participants with 1+ contact recruited.) | 24; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities (In a stepped-wedge trial, enrollment is zero by design for certain sequences in certain periods.) | 53; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities (In a stepped-wedge trial, enrollment is zero by design for certain sequences in certain periods.) | 31; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities (In a stepped-wedge trial, enrollment is zero by design for certain sequences in certain periods.) | 35; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities (In a stepped-wedge trial, enrollment is zero by design for certain sequences in certain periods.) | 22; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities (In a stepped-wedge trial, enrollment is zero by design for certain sequences in certain periods.) | 51; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities (In a stepped-wedge trial, enrollment is zero by design for certain sequences in certain periods.)
Close Contacts (Close contacts of index participants who were screened for TB.) | 61; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities (In a stepped-wedge trial, enrollment is zero by design for certain sequences in certain periods.) | 244; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities (In a stepped-wedge trial, enrollment is zero by design for certain sequences in certain periods.) | 80; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities (In a stepped-wedge trial, enrollment is zero by design for certain sequences in certain periods.) | 99; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities (In a stepped-wedge trial, enrollment is zero by design for certain sequences in certain periods.) | 88; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities (In a stepped-wedge trial, enrollment is zero by design for certain sequences in certain periods.) | 125; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities (In a stepped-wedge trial, enrollment is zero by design for certain sequences in certain periods.)
Completed | 85; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities (In a stepped-wedge trial, enrollment is zero by design for certain sequences in certain periods.) | 297; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities (In a stepped-wedge trial, enrollment is zero by design for certain sequences in certain periods.) | 111; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities (In a stepped-wedge trial, enrollment is zero by design for certain sequences in certain periods.) | 134; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities (In a stepped-wedge trial, enrollment is zero by design for certain sequences in certain periods.) | 110; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities (In a stepped-wedge trial, enrollment is zero by design for certain sequences in certain periods.) | 176; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities (In a stepped-wedge trial, enrollment is zero by design for certain sequences in certain periods.)
Not Completed | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities
Period: Period 2 (Weeks 9-16)
Arm/Group | Standard Contact Investigation [Control]: Sequence 1 [2 Health Facilities] | User-centered Contact Investigation [Intervention]: Sequence 1 [2 Health Facilities] | Standard Contact Investigation [Control]: Sequence 2 [2 Health Facilities] | User-centered Contact Investigation [Intervention]: Sequence 2 [2 Health Facilities] | Standard Contact Investigation [Control]: Sequence 3 [2 Health Facilities] | User-centered Contact Investigation [Intervention]: Sequence 3 [2 Health Facilities] | Standard Contact Investigation [Control]: Sequence 4 [2 Health Facilities] | User-centered Contact Investigation [Intervention]: Sequence 4 [2 Health Facilities] | Standard Contact Investigation [Control]: Sequence 5 [2 Health Facilities] | User-centered Contact Investigation [Intervention]: Sequence 5 [2 Health Facilities] | Standard Contact Investigation [Control]: Sequence 6 [2 Health Facilities] | User-centered Contact Investigation [Intervention]: Sequence 6 [2 Health Facilities]
Started | 0; 0 Pairs of Health Facilities (In a stepped-wedge trial with a cross-sectional outcome, participants are included in one period only.) | 0; 0 Pairs of Health Facilities | 353; 1 Pairs of Health Facilities (In a stepped-wedge trial with a cross-sectional outcome, participants are included in one period only.) | 0; 0 Pairs of Health Facilities | 167; 1 Pairs of Health Facilities (In a stepped-wedge trial with a cross-sectional outcome, participants are included in one period only.) | 0; 0 Pairs of Health Facilities | 98; 1 Pairs of Health Facilities (In a stepped-wedge trial with a cross-sectional outcome, participants are included in one period only.) | 0; 0 Pairs of Health Facilities | 124; 1 Pairs of Health Facilities (In a stepped-wedge trial with a cross-sectional outcome, participants are included in one period only.) | 0; 0 Pairs of Health Facilities | 266; 1 Pairs of Health Facilities (In a stepped-wedge trial with a cross-sectional outcome, participants are included in one period only.) | 0; 0 Pairs of Health Facilities
Index Participants | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 64; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 43; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 30; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 25; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 69; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities
Close Contacts | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 289; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 124; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 68; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 99; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 197; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities
Completed | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 353; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 167; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 98; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 124; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 266; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities
Not Completed | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities
Period: Period 3 (Weeks 17-24)
Arm/Group | Standard Contact Investigation [Control]: Sequence 1 [2 Health Facilities] | User-centered Contact Investigation [Intervention]: Sequence 1 [2 Health Facilities] | Standard Contact Investigation [Control]: Sequence 2 [2 Health Facilities] | User-centered Contact Investigation [Intervention]: Sequence 2 [2 Health Facilities] | Standard Contact Investigation [Control]: Sequence 3 [2 Health Facilities] | User-centered Contact Investigation [Intervention]: Sequence 3 [2 Health Facilities] | Standard Contact Investigation [Control]: Sequence 4 [2 Health Facilities] | User-centered Contact Investigation [Intervention]: Sequence 4 [2 Health Facilities] | Standard Contact Investigation [Control]: Sequence 5 [2 Health Facilities] | User-centered Contact Investigation [Intervention]: Sequence 5 [2 Health Facilities] | Standard Contact Investigation [Control]: Sequence 6 [2 Health Facilities] | User-centered Contact Investigation [Intervention]: Sequence 6 [2 Health Facilities]
Started | 0; 0 Pairs of Health Facilities | 304; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 238; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 73; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 155; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 217; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities
Index Participants | 0; 0 Pairs of Health Facilities | 53; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 49; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 20; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 29; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 55; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities
Close Contacts | 0; 0 Pairs of Health Facilities | 251; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 189; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 53; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 126; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 162; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities
Completed | 0; 0 Pairs of Health Facilities | 304; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 238; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 73; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 155; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 217; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities
Not Completed | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities
Period: Period 4 (Weeks 25-32)
Arm/Group | Standard Contact Investigation [Control]: Sequence 1 [2 Health Facilities] | User-centered Contact Investigation [Intervention]: Sequence 1 [2 Health Facilities] | Standard Contact Investigation [Control]: Sequence 2 [2 Health Facilities] | User-centered Contact Investigation [Intervention]: Sequence 2 [2 Health Facilities] | Standard Contact Investigation [Control]: Sequence 3 [2 Health Facilities] | User-centered Contact Investigation [Intervention]: Sequence 3 [2 Health Facilities] | Standard Contact Investigation [Control]: Sequence 4 [2 Health Facilities] | User-centered Contact Investigation [Intervention]: Sequence 4 [2 Health Facilities] | Standard Contact Investigation [Control]: Sequence 5 [2 Health Facilities] | User-centered Contact Investigation [Intervention]: Sequence 5 [2 Health Facilities] | Standard Contact Investigation [Control]: Sequence 6 [2 Health Facilities] | User-centered Contact Investigation [Intervention]: Sequence 6 [2 Health Facilities]
Started | 0; 0 Pairs of Health Facilities | 311; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 495; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 166; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 105; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 227; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities
Index Participants | 0; 0 Pairs of Health Facilities | 62; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 69; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 48; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 17; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 55; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities
Close Contacts | 0; 0 Pairs of Health Facilities | 249; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 426; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 118; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 88; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 172; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities
Completed | 0; 0 Pairs of Health Facilities | 311; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 495; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 166; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 105; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 227; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities
Not Completed | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities
Period: Period 5 (Weeks 33-40)
Arm/Group | Standard Contact Investigation [Control]: Sequence 1 [2 Health Facilities] | User-centered Contact Investigation [Intervention]: Sequence 1 [2 Health Facilities] | Standard Contact Investigation [Control]: Sequence 2 [2 Health Facilities] | User-centered Contact Investigation [Intervention]: Sequence 2 [2 Health Facilities] | Standard Contact Investigation [Control]: Sequence 3 [2 Health Facilities] | User-centered Contact Investigation [Intervention]: Sequence 3 [2 Health Facilities] | Standard Contact Investigation [Control]: Sequence 4 [2 Health Facilities] | User-centered Contact Investigation [Intervention]: Sequence 4 [2 Health Facilities] | Standard Contact Investigation [Control]: Sequence 5 [2 Health Facilities] | User-centered Contact Investigation [Intervention]: Sequence 5 [2 Health Facilities] | Standard Contact Investigation [Control]: Sequence 6 [2 Health Facilities] | User-centered Contact Investigation [Intervention]: Sequence 6 [2 Health Facilities]
Started | 0; 0 Pairs of Health Facilities | 247; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 385; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 563; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 175; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 163; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities
Index Participants | 0; 0 Pairs of Health Facilities | 38; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 43; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 71; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 29; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 40; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities
Close Contacts | 0; 0 Pairs of Health Facilities | 209; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 342; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 492; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 146; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 123; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities
Completed | 0; 0 Pairs of Health Facilities | 247; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 385; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 563; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 175; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 163; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities
Not Completed | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities
Period: Period 6 (Week 41-48)
Arm/Group | Standard Contact Investigation [Control]: Sequence 1 [2 Health Facilities] | User-centered Contact Investigation [Intervention]: Sequence 1 [2 Health Facilities] | Standard Contact Investigation [Control]: Sequence 2 [2 Health Facilities] | User-centered Contact Investigation [Intervention]: Sequence 2 [2 Health Facilities] | Standard Contact Investigation [Control]: Sequence 3 [2 Health Facilities] | User-centered Contact Investigation [Intervention]: Sequence 3 [2 Health Facilities] | Standard Contact Investigation [Control]: Sequence 4 [2 Health Facilities] | User-centered Contact Investigation [Intervention]: Sequence 4 [2 Health Facilities] | Standard Contact Investigation [Control]: Sequence 5 [2 Health Facilities] | User-centered Contact Investigation [Intervention]: Sequence 5 [2 Health Facilities] | Standard Contact Investigation [Control]: Sequence 6 [2 Health Facilities] | User-centered Contact Investigation [Intervention]: Sequence 6 [2 Health Facilities]
Started | 0; 0 Pairs of Health Facilities | 193; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 414; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 395; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 241; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 277; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities
Index Participants | 0; 0 Pairs of Health Facilities | 38; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 56; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 50; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 42; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 54; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities
Close Contacts | 0; 0 Pairs of Health Facilities | 155; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 358; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 345; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 199; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 223; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities
Completed | 0; 0 Pairs of Health Facilities | 193; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 414; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 395; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 241; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 277; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities
Not Completed | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities
Period: Period 7 (Weeks 49-56)
Arm/Group | Standard Contact Investigation [Control]: Sequence 1 [2 Health Facilities] | User-centered Contact Investigation [Intervention]: Sequence 1 [2 Health Facilities] | Standard Contact Investigation [Control]: Sequence 2 [2 Health Facilities] | User-centered Contact Investigation [Intervention]: Sequence 2 [2 Health Facilities] | Standard Contact Investigation [Control]: Sequence 3 [2 Health Facilities] | User-centered Contact Investigation [Intervention]: Sequence 3 [2 Health Facilities] | Standard Contact Investigation [Control]: Sequence 4 [2 Health Facilities] | User-centered Contact Investigation [Intervention]: Sequence 4 [2 Health Facilities] | Standard Contact Investigation [Control]: Sequence 5 [2 Health Facilities] | User-centered Contact Investigation [Intervention]: Sequence 5 [2 Health Facilities] | Standard Contact Investigation [Control]: Sequence 6 [2 Health Facilities] | User-centered Contact Investigation [Intervention]: Sequence 6 [2 Health Facilities]
Started | 0; 0 Pairs of Health Facilities | 273; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 367; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 257; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 283; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 216; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities
Index Participants | 0; 0 Pairs of Health Facilities | 46; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 50; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 37; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 53; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 29; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities
Close Contacts | 0; 0 Pairs of Health Facilities | 227; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 317; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 220; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 230; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 187; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities
Completed | 0; 0 Pairs of Health Facilities | 273; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 367; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 257; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 283; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 216; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities
Not Completed | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities
Period: Period 8 (Weeks 57-64)
Arm/Group | Standard Contact Investigation [Control]: Sequence 1 [2 Health Facilities] | User-centered Contact Investigation [Intervention]: Sequence 1 [2 Health Facilities] | Standard Contact Investigation [Control]: Sequence 2 [2 Health Facilities] | User-centered Contact Investigation [Intervention]: Sequence 2 [2 Health Facilities] | Standard Contact Investigation [Control]: Sequence 3 [2 Health Facilities] | User-centered Contact Investigation [Intervention]: Sequence 3 [2 Health Facilities] | Standard Contact Investigation [Control]: Sequence 4 [2 Health Facilities] | User-centered Contact Investigation [Intervention]: Sequence 4 [2 Health Facilities] | Standard Contact Investigation [Control]: Sequence 5 [2 Health Facilities] | User-centered Contact Investigation [Intervention]: Sequence 5 [2 Health Facilities] | Standard Contact Investigation [Control]: Sequence 6 [2 Health Facilities] | User-centered Contact Investigation [Intervention]: Sequence 6 [2 Health Facilities]
Started | 0; 0 Pairs of Health Facilities | 188; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 322; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 448; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 317; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 227; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 314; 1 Pairs of Health Facilities
Index Participants | 0; 0 Pairs of Health Facilities | 36; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 41; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 48; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 61; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 35; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 41; 1 Pairs of Health Facilities
Close Contacts | 0; 0 Pairs of Health Facilities | 152; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 281; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 400; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 256; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 192; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 273; 1 Pairs of Health Facilities
Completed | 0; 0 Pairs of Health Facilities | 188; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 322; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 448; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 317; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 227; 1 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 314; 1 Pairs of Health Facilities
Not Completed | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities | 0; 0 Pairs of Health Facilities

BASELINE CHARACTERISTICS:
Population: Provided are baseline characteristics for all that participated- both index and household contact participants.
Groups:
- Standard Contact Investigation: Index Participants; Standard Contact Investigation: Household Contacts: Standard contact investigation consists of 1) evidence-based procedures for TB contact investigation, introduced with 2) a standard implementation strategy.
  Standard contact investigation:
  Once an eligible TB patient agrees to participate, CHWs will visit the patient to assess the eligibility of close contacts to participate.
  For eligible contacts who agree to participate, the CHW will perform TB symptom screening and arrange subsequent microbiologic, clinical, and/or radiographic evaluation. Those screening TB symptom-positive will be asked to expectorate a sputum sample, unless under age 5. If under age 5 or unable to produce sputum, contacts will be referred to the health centre for evaluation. A CHW will transport sputum samples to the health-centre laboratory for microbiologic evaluation and later report the test results back to the contact.
  Standard Implementation Strategy:
  CHWs at all sites will receive the standard TB program training on TB contact investigation and supportive supervision from the on-site National TB Program focal person.
- User-centered Contact Investigation: Index Participants; User-centered Contact Investigation: Household Contacts: User-centered Contact Investigation includes 4 client-facing adaptations of standard contact investigation and 3 CHW-facing implementation strategies Client-centered adaptations of contact investigation delivered as a branded package called Tuli Wamu Nawe: Four novel tools TB education pamphlet to help index TB persons disclose the need for TB screening to close contacts.
  Contact identification algorithm to help CHWs and index TB persons accurately enumerate contacts.
  Sputum collection video to instruct contacts to expectorate good-quality sputum.
  Community Health Riders to transport CHWs, index persons with TB, and contacts by motorcycle taxi, and collect and transport sputum.
  CHW-centered Implementation Strategy: Three components Weekly CHW meetings to create communities of practice (CoP), which consist of professionals organized for peer support and systematic learning.
  Audit and feedback reports on contact investigation performance indicators delivered weekly (individual CHW) and monthly (health facility).
  A group-chat application to facilitate peer support among CHWs.
- Total: Total of all reporting groups
Arm/Group | Standard Contact Investigation: Index Participants | Standard Contact Investigation: Household Contacts | User-centered Contact Investigation: Index Participants | User-centered Contact Investigation: Household Contacts | Total
Number analyzed (Participants) | 843 | 2874 | 999 | 5761 | 10477
Age, Customized [Count of Participants; unit: Participants]
  <5 years | 81 | 310 | 63 | 648 | 1102
  5-14 years | 51 | 808 | 49 | 1603 | 2511
  ≥15 years | 711 | 1756 | 887 | 3510 | 6864
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 379 | 1591 | 415 | 2987 | 5372
  Male | 464 | 1283 | 584 | 2774 | 5105
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 843 | 2874 | 999 | 5761 | 10477
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 843 | 2874 | 999 | 5761 | 10477
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Uganda | 843 | 2874 | 999 | 5761 | 10477
Person living with HIV [Number; unit: participants] | 343 | 142 | 461 | 235 | 1181

OUTCOME MEASURES:

1. Primary Outcome: Completion of TB Evaluation
Description: The percentage of participants (close contacts) who are experiencing TB symptoms who complete TB evaluation within 60 days of the TB patient's treatment initiation date
Time Frame: 60 days
Population: Only those who screened positive for symptoms of TB are included in this analysis
Measure: Count of Participants; unit: Participants
Groups:
- Enhanced Contact Investigation Intervention Period: The enhanced contact investigation strategy includes 4 implementation facilitation tools and 3 continuous quality improvement techniques delivered as a branded package. Implementation tools include 1) a TB education pamphlet, 2) a contact identification algorithm, 3) an instructional video on sputum collection, and 4) community health riders who transport clients, community health workers, and sputum samples by motorcycle. The continuous quality improvement techniques delivered as the community of practice package include 1) community of practice meetings, 2) audit and feedback reports and 3) a group chat application.
  User-Centered Implementation Strategy: 1) 4 participant-facing components: 1a) TB education pamphlet helps index TB persons disclose the need for household screening to contacts. 1b) Contact identification algorithm helps CHWs and index TB persons accurately enumerate contacts. 1c) Sputum collection video instructs contacts to expectorate good-quality sputum. 1d) Community Health Riders transport CHWs, index persons with TB, and contacts by motorcycle taxi, and collect and transport sputum.
  2) 3 community health-worker-facing components: a) Weekly CHW meetings create communities of practice (CoP), professionals organized for peer support and systematic learning. 2b) Audit and feedback reports on contact investigation performance indicators weekly (individual CHW) and monthly (health facility). 2c) A group-chat application facilitates peer support among CHWs.
Arm/Group | Standard Implementation Strategy Period | Enhanced Contact Investigation Intervention Period
Number analyzed (Participants) | 560 | 1329
Participants | 266 | 1144
Statistical Analysis 1: Comparison: Standard Implementation Strategy Period vs Enhanced Contact Investigation Intervention Period; Test type: Other; p < 0.001, Mixed Models Analysis; Mixed-effects Poisson model adjusting for time and group level (paired health centres, based on randomization) cluster; Incidence rate ratio = 1.84, 95% CI 2-sided [1.62 to 2.09]

2. Secondary Outcome: TB Yield (Diagnosis and Treatment Initiation)
Description: The difference between study periods in percentage of contacts diagnosed with active TB and initiated on treatment within 60 days of the TB patient's treatment initiation
Time Frame: 60 days
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Implementation Strategy Period | Enhanced Contact Investigation Intervention Period
Number analyzed (Participants) | 2874 | 5761
Participants | 36 | 187
Statistical Analysis 1: Comparison: Standard Implementation Strategy Period vs Enhanced Contact Investigation Intervention Period; Test type: Other; p = 0.002, Mixed Models Analysis; Mixed-effects Poisson model adjusting for time and group level (paired health centres, based on randomization) cluster; Incidence Rate Ratio = 7.46, 95% CI 2-sided [2.06 to 26.95]

3. Secondary Outcome: Initiation of TB Preventative Therapy
Description: The difference between study periods in percentage of contacts initiating TB preventative therapy (TPT) within 60 days of the TB patient's treatment initiation
Time Frame: 60 days
Population: Only those eligible for TPT are included in this analysis. Those that have been newly diagnosed with TB, regardless of treatment status, are not eligible for TPT and are therefore excluded from this analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Implementation Strategy Period | Enhanced Contact Investigation Intervention Period
Number analyzed (Participants) | 2829 | 5560
Participants | 122 | 264
Statistical Analysis 1: Comparison: Standard Implementation Strategy Period vs Enhanced Contact Investigation Intervention Period; Test type: Other; p = 0.50, Mixed Models Analysis; Mixed effects poisson model adjusting for time and group (paired healthcentres, based on randomization); Incidence Rate Ratio = 1.25, 95% CI 2-sided [0.65 to 2.42]

4. Secondary Outcome: Number of Contacts Diagnosed With Active TB
Description: The difference between study periods in counts of the number of contacts diagnosed with active TB
Time Frame: 60 days
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Implementation Strategy Period | Enhanced Contact Investigation Intervention Period
Number analyzed (Participants) | 2874 | 5761
Participants | 45 | 201

5. Secondary Outcome: Number of Contacts Initiating TB Preventative Therapy
Description: The difference between study periods in counts of the number of contacts initiating TPT
Time Frame: 60 days
Population: This outcome is only for those eligible to initiate TPT. Those who have been newly diagnosed, regardless of treatment status, are not eligible for TPT and are therefore excluded from this outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Implementation Strategy Period | Enhanced Contact Investigation Intervention Period
Number analyzed (Participants) | 2829 | 5560
Participants | 122 | 264

6. Secondary Outcome: TB Yield (All Contacts)
Description: The difference between study periods in percentage of all TB cases among contacts
Time Frame: 60 days
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Implementation Strategy Period | Enhanced Contact Investigation Intervention Period
Number analyzed (Participants) | 2874 | 5761
Participants | 45 | 201
Statistical Analysis 1: Comparison: Standard Implementation Strategy Period vs Enhanced Contact Investigation Intervention Period; Test type: Other; p < 0.001, Mixed Models Analysis; Mixed-effects Poisson model adjusting for time and group level (paired health centres, based on randomization) cluster; Incidence Rate Ratio = 4.75, 95% CI 2-sided [2.07 to 10.91]

ADVERSE EVENTS:
Time Frame: 60 days
Description: All-Cause Mortality was not collected.
Groups:
- Standard Contact Investigation [Control]: Sequence 1 [2 Health Facilities]: Cluster 1: 8 weeks of standard, then 8 weeks of transition, then 48 weeks of user-centered
  ----------------- Standard contact investigation consists of 1) evidence-based procedures for TB contact investigation, introduced with 2) a standard implementation strategy.
  1. Standard contact investigation:
     1. Once an eligible TB patient agrees to participate, CHWs will visit the patient to assess the eligibility of close contacts to participate.
     2. For eligible contacts who agree to participate, the CHW will perform TB symptom screening and arrange subsequent microbiologic, clinical, and/or radiographic evaluation.
     3. Those screening TB symptom-positive will be asked to expectorate a sputum sample, unless under age 5. If under age 5 or unable to produce sputum, contacts will be referred to the health centre for evaluation. A CHW will transport sputum samples to the health-centre laboratory for microbiologic evaluation and later report the test results back to the contact.
  2. Standard Implementation Strategy:
  CHWs at all sites will receive the standard TB program training on TB contact investigation and supportive supervision from the on-site National TB Program focal person.
- Standard Contact Investigation [Control]: Sequence 2 [2 Health Facilities]: Cluster 2: 16 weeks of standard, then 8 weeks of transition, then 40 weeks of user-centered
  ----------------- Standard contact investigation consists of 1) evidence-based procedures for TB contact investigation, introduced with 2) a standard implementation strategy.
  1. Standard contact investigation:
     1. Once an eligible TB patient agrees to participate, CHWs will visit the patient to assess the eligibility of close contacts to participate.
     2. For eligible contacts who agree to participate, the CHW will perform TB symptom screening and arrange subsequent microbiologic, clinical, and/or radiographic evaluation.
     3. Those screening TB symptom-positive will be asked to expectorate a sputum sample, unless under age 5. If under age 5 or unable to produce sputum, contacts will be referred to the health centre for evaluation. A CHW will transport sputum samples to the health-centre laboratory for microbiologic evaluation and later report the test results back to the contact.
  2. Standard Implementation Strategy:
  CHWs at all sites will receive the standard TB program training on TB contact investigation and supportive supervision from the on-site National TB Program focal person.
- Standard Contact Investigation [Control]: Sequence 3 [2 Health Facilities]: Cluster 3: 24 weeks of standard, then 8 weeks of transition, then 32 weeks of user-centered
  ----------------- Standard contact investigation consists of 1) evidence-based procedures for TB contact investigation, introduced with 2) a standard implementation strategy.
  1. Standard contact investigation:
     1. Once an eligible TB patient agrees to participate, CHWs will visit the patient to assess the eligibility of close contacts to participate.
     2. For eligible contacts who agree to participate, the CHW will perform TB symptom screening and arrange subsequent microbiologic, clinical, and/or radiographic evaluation.
     3. Those screening TB symptom-positive will be asked to expectorate a sputum sample, unless under age 5. If under age 5 or unable to produce sputum, contacts will be referred to the health centre for evaluation. A CHW will transport sputum samples to the health-centre laboratory for microbiologic evaluation and later report the test results back to the contact.
  2. Standard Implementation Strategy:
  CHWs at all sites will receive the standard TB program training on TB contact investigation and supportive supervision from the on-site National TB Program focal person.
- Standard Contact Investigation [Control]: Sequence 4 [2 Health Facilities]: Cluster 4: 32 weeks of standard, then 8 weeks of transition, then 24 weeks of user-centered
  ----------------- Standard contact investigation consists of 1) evidence-based procedures for TB contact investigation, introduced with 2) a standard implementation strategy.
  1. Standard contact investigation:
     1. Once an eligible TB patient agrees to participate, CHWs will visit the patient to assess the eligibility of close contacts to participate.
     2. For eligible contacts who agree to participate, the CHW will perform TB symptom screening and arrange subsequent microbiologic, clinical, and/or radiographic evaluation.
     3. Those screening TB symptom-positive will be asked to expectorate a sputum sample, unless under age 5. If under age 5 or unable to produce sputum, contacts will be referred to the health centre for evaluation. A CHW will transport sputum samples to the health-centre laboratory for microbiologic evaluation and later report the test results back to the contact.
  2. Standard Implementation Strategy:
  CHWs at all sites will receive the standard TB program training on TB contact investigation and supportive supervision from the on-site National TB Program focal person.
- Standard Contact Investigation [Control]: Sequence 5 [2 Health Facilities]: Cluster 5: 40 weeks of standard, then 8 weeks of transition, then 16 weeks of user-centered
  ----------------- Standard contact investigation consists of 1) evidence-based procedures for TB contact investigation, introduced with 2) a standard implementation strategy.
  1. Standard contact investigation:
     1. Once an eligible TB patient agrees to participate, CHWs will visit the patient to assess the eligibility of close contacts to participate.
     2. For eligible contacts who agree to participate, the CHW will perform TB symptom screening and arrange subsequent microbiologic, clinical, and/or radiographic evaluation.
     3. Those screening TB symptom-positive will be asked to expectorate a sputum sample, unless under age 5. If under age 5 or unable to produce sputum, contacts will be referred to the health centre for evaluation. A CHW will transport sputum samples to the health-centre laboratory for microbiologic evaluation and later report the test results back to the contact.
  2. Standard Implementation Strategy:
  CHWs at all sites will receive the standard TB program training on TB contact investigation and supportive supervision from the on-site National TB Program focal person.
- Standard Contact Investigation [Control]: Sequence 6 [2 Health Facilities]: Cluster 6: 48 weeks of standard, then 8 weeks of transition, then 8 weeks of user-centered
  ----------------- Standard contact investigation consists of 1) evidence-based procedures for TB contact investigation, introduced with 2) a standard implementation strategy.
  1. Standard contact investigation:
     1. Once an eligible TB patient agrees to participate, CHWs will visit the patient to assess the eligibility of close contacts to participate.
     2. For eligible contacts who agree to participate, the CHW will perform TB symptom screening and arrange subsequent microbiologic, clinical, and/or radiographic evaluation.
     3. Those screening TB symptom-positive will be asked to expectorate a sputum sample, unless under age 5. If under age 5 or unable to produce sputum, contacts will be referred to the health centre for evaluation. A CHW will transport sputum samples to the health-centre laboratory for microbiologic evaluation and later report the test results back to the contact.
  2. Standard Implementation Strategy:
  CHWs at all sites will receive the standard TB program training on TB contact investigation and supportive supervision from the on-site National TB Program focal person.
Arm/Group | Standard Contact Investigation [Control]: Sequence 1 [2 Health Facilities] | User-centered Contact Investigation [Intervention]: Sequence 1 [2 Health Facilities] | Standard Contact Investigation [Control]: Sequence 2 [2 Health Facilities] | User-centered Contact Investigation [Intervention]: Sequence 2 [2 Health Facilities] | Standard Contact Investigation [Control]: Sequence 3 [2 Health Facilities] | User-centered Contact Investigation [Intervention]: Sequence 3 [2 Health Facilities] | Standard Contact Investigation [Control]: Sequence 4 [2 Health Facilities] | User-centered Contact Investigation [Intervention]: Sequence 4 [2 Health Facilities] | Standard Contact Investigation [Control]: Sequence 5 [2 Health Facilities] | User-centered Contact Investigation [Intervention]: Sequence 5 [2 Health Facilities] | Standard Contact Investigation [Control]: Sequence 6 [2 Health Facilities] | User-centered Contact Investigation [Intervention]: Sequence 6 [2 Health Facilities]
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/85 | 0/1516 | 0/650 | 0/1983 | 0/516 | 0/1663 | 0/471 | 0/841 | 0/669 | 0/443 | 0/1326 | 0/314
Other Adverse Events (participants affected / at risk) | 0/85 | 0/1516 | 0/650 | 0/1983 | 0/516 | 0/1663 | 0/471 | 0/841 | 0/669 | 0/443 | 0/1326 | 0/314

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2022-09-12): https://cdn.clinicaltrials.gov/large-docs/48/NCT05640648/Prot_002.pdf
  • Statistical Analysis Plan (2023-05-02): https://cdn.clinicaltrials.gov/large-docs/48/NCT05640648/SAP_003.pdf
  • Informed Consent Form (2022-09-12): https://cdn.clinicaltrials.gov/large-docs/48/NCT05640648/ICF_004.pdf